CLINICAL TRIAL: NCT03515941
Title: A Pilot Study in Gastric Cancer of Assignment to Postoperative Chemoradiation or Chemotherapy Based Upon Surgical Lymph Node Assessment After Preoperative Chemotherapy, With Gene Assay as Correlate of Biologic Response
Brief Title: Postoperative Chemoradiation or Chemotherapy After Preoperative Chemotherapy for Gastric Cancers
Acronym: GABLE
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: The PI has decided to close the study due to the outdated study design.
Sponsor: Tannaz Armaghany (Other)
Responsible Party: Sponsor-Investigator, Tannaz Armaghany, Assistant Professor of Medicine - Hematology and Oncology, Baylor College of Medicine
Organization: Baylor College of Medicine (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-40682
Record Dates: First submitted 2018-04-24; First posted 2018-05-04 (Actual); Results first posted 2020-10-12 (Actual); Last update posted 2020-10-12 (Actual); Status verified 2020-10

CONDITIONS: Gastrointestinal Cancer
Keywords: chemotherapy; chemoradiation
MeSH Terms: conditions — Gastrointestinal Neoplasms | interventions — Oxaliplatin; Capecitabine; Leucovorin; Fluorouracil; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1: Adjuvant Chemotherapy (Experimental): Three cycles of chemo with CAPEOX (Oxaliplatin:130 mg/m2 by IV and Capecitabine: 625 or 1000 mg/m2 by PO (BID) on 21 day-cycle or FOLFOX (Oxaliplatin:85 mg/m2 by IV, Leucovorin:400 mg/m2 by IV,5-fluorouracil: 400 mg/m2 and 2400 mg/m2 by IV) on 14 day-cycle
  Interventions: Drug: Oxaliplatin; Drug: Capecitabine; Drug: Leucovorin; Drug: 5-fluorouracil
- Arm 2: Adjuvant Chemoradiation (Experimental): Three cycles of chemo with Capecitabine: 750 mg/m2 by PO BID on days 1-14 of a 28 day-cycle or 5-fluorouracil (Leucovorin:400 mg/m2 by IV,5-fluorouracil: 400 mg/m2 and 1200 mg/m2 by IV) on days 1 and 15 of a 28 day cycle After 1st chemo cycle above, chemoradiation for 5 weeks with 45 Gy in 1.8 Gy/fraction, 5 days a week, to the entire gastric bed (including anastomosis) and draining lymph nodes, and a single agent fluoropyrimidine, either capecitabine or 5-fluorouracil After 5 weeks chemoradiation, 2 cycles of chemo as described above.
  Interventions: Drug: Capecitabine; Drug: Leucovorin; Drug: 5-fluorouracil; Radiation: radiation

INTERVENTIONS:
Drug: Oxaliplatin — 130 mg/m2 by IV (Arm 1)
  Other Names: Eloxatin
  Arms: Arm 1: Adjuvant Chemotherapy
Drug: Capecitabine — 625 mg/m2 (Arm 1), 1000 mg/m2 (Arm 1), 750 mg/m2 by PO (Arm 2)
  Other Names: Xeloda
Drug: Leucovorin — 400 mg/m2 by IV (Arm 1 & Arm 2)
  Other Names: Wellcovorin
Drug: 5-fluorouracil — 400, 2400 mg/m2 by IV (Arm 1), 400,1200 mg/m2 by IV (Arm 2)
  Other Names: Adrucil
Radiation: radiation — 45 Gy in 1.8 Gy/fraction
  Arms: Arm 2: Adjuvant Chemoradiation

SUMMARY:
This is an open-label, stratified, two arm design. All patients receive same initial standard preoperative chemotherapy and surgical resection. Patients will then be assigned to either standard postoperative chemotherapy if node negative at surgery or standard postoperative chemoradiation if node positive at surgery.

The primary objective of this study is to determine the feasibility of patients enrolling and receiving either postoperative chemoradiation or chemotherapy alone, based upon nodal status at surgery, following preoperative chemotherapy.

The secondary Objectives is to evaluate the rate of cancer recurrence in patients assigned to treatment based upon node status. To explore the potential correlation between changes in expression of a pre-specified panel of genes identified as relevant to gastrointestinal cancers in response to preoperative chemotherapy, using presence of nodal involvement at time of surgery as an indicator of response.

DETAILED DESCRIPTION:
Gastric adenocarcinoma, also known as stomach cancer, is a global health problem. While surgical resection remains the only curative option for patients who develop this disease, because of its aggressive nature and high recurrence rates, all but the lowest stages of gastric cancer require additional, adjuvant therapy in addition to surgery. Currently, two competing standards exist for the adjuvant management of gastric cancer: peri-operative chemotherapy (based upon the MAGIC study), and postoperative combination chemoradiation therapy (based upon the MacDonald Intergroup study). These two standards were arrived at based upon two separate trials that did not directly compare the two approaches, and thus either approach is considered acceptable. Several modifications to the chemotherapy used in the peri-operative approach have been studied and are now accepted as standard as well. Selection oftentimes derives from physician preference and tumor characteristics such as symptoms or nodal stage, and a clear guideline for when to select one adjuvant approach over the other is lacking.

Currently, analysis of patient outcomes from the large, randomized phase III CRITICS trial is ongoing, and will attempt to answer if one approach is clearly favored. Patients enrolled in the CRITICS trial all received preoperative chemotherapy and standardized surgical resection. Patients were then randomized to receive either chemotherapy or chemoradiation therapies postoperatively. Enrollment is closed for the CRITICS trial; preliminary data suggest that neither arm of postoperative treatment is superior. These early data support what practitioners have long suspected, which is that no one adjuvant standard is universally superior, but that tumors from different patients and with different characteristics will respond better to different adjuvant approaches.

Unfortunately, knowing which tumors will respond better to which therapy remains unpredictable. Certain clinical features can help clinicians to make a recommendation for their adjuvant approach. For example, patients who have tumors that are symptomatic, such as with bleeding or gastric obstruction, are less likely to tolerate several months of surgical delay while chemotherapy is administered preoperatively, and thus will typically be offered upfront surgery, followed by adjuvant chemoradiation. For most patients, however, the administration of systemic therapy prior to surgery as a part of a perioperative approach is recommended. This approach is favored because of the local control and reduction in tumor that can result prior to surgery, which is thought to lead to better outcomes in the long term.

However, not all patients will experience a response to preoperative chemotherapy. In those patients whose tumors are found at surgery to remain advanced, with nodal involvement, despite preoperative chemotherapy, long-term outcomes have been shown to be poorer than those whose tumors responded well, with the absence of nodal involvement upon dissection. These data are based upon the retrospective analysis of those patients who were enrolled in the original MAGIC study. Approximately 75% of tumors were found to be in the category of having nodes involved with cancer at resection despite preoperative chemotherapy. Thus, for this majority of patients with gastric cancer who have an inadequate response to preoperative chemotherapy (i.e., who remain node-positive at surgery), an alternative approach to their postoperative adjuvant treatment rather than mere completion of postoperative chemotherapy is apparently necessary.

One reasonable alternative for the management of patients who remain node positive at surgery could be to incorporate radiation into their postoperative adjuvant treatment. There is some evidence for this approach, coming from the South Korean ARTIST trial. In the ARTIST trial, patients who underwent gastrectomy for stomach cancer randomly received either post-operative chemotherapy or chemoradiation therapy. Although no overall survival benefit was seen overall in the ARTIST study, in subset analysis, node positive patients had a significant improvement in disease-free survival with adjuvant chemoradiotherapy versus adjuvant chemotherapy alone.

The disparity in tumor responses to preoperative chemotherapy supports biologic heterogeneity of these tumors. Understanding these biologic differences would be invaluable to the future therapeutic direction of their management. These differences are likely complex, existing as baseline genetic characteristics at diagnosis but also as dynamic changes in these characteristics in response to chemotherapy. Identifying these characteristics could allow clinicians to determine which patients' tumors are unlikely to respond to therapy upfront or how to modify ongoing therapy in response to tumor response and evolution as therapy is administered. Knowing that tumor nodal response to preoperative chemotherapy is a surrogate for outcomes in these patients can provide an important comparator for groups of gene expression and evolution.

Recent work into the characterization of gastric adenocarcinoma suggests that four distinct molecular subtypes exist. These subtypes are characterized as Epstein-Barr virus positive, microsatellite unstable, genomically stable, and chromosome instable. Determination of the genetic features giving rise to each category is based upon analysis of virgin tumor samples, and thus does not consider variations that arise in response to treatment. Nevertheless, each subtype is characterized by the expression or mutation of specific genes or gene categories that can be profiled through routine analysis. Correlating these gene expressions to clinical nodal responses to chemotherapy could potentially offer insights into the biomarker driven determination of adjuvant treatment selection in gastric cancer. Additionally, monitoring these gene expression levels in response to therapy and making similar correlates could provide valuable information into the adaption of adjuvant therapy to the tumor's response to treatment in real time.

The genes associated with these four proposed subtypes of gastric cancer are by no means exhaustive, however, and the expression or alteration of other genes may yield further predictive and therapeutic information for the adjuvant treatment of these cancers. Casting a wider net is increasingly easy to accomplish, with the advent of genomic profiling of tumors. Particularly in the case of profiles that assess for expression of targetable genes, the ability to assess or monitor for their expression as they relate to chemotherapy response could have important implications for being able to incorporate the therapies into the adjuvant treatment process at critical junctures in the treatment sequence.

ELIGIBILITY:
Inclusion Criteria:

1. Must have pathologically-proven adenocarcinoma of the stomach or gastroesophageal (GE)-junction, stage M0, as established by both imaging and surgical pathologic staging.

   Imaging: Clinical stage of M0 will be established by either CT (chest with contrast and abdomen/pelvis with and without contrast), or CT/PET (positron emission tomography) (skull base to mid-thigh). This is standard post-surgery imaging.

   Surgery: Surgical pathologic staging must be M0.
2. Must have completed 3 cycles of neo-adjuvant chemotherapy. Either CAPEOX or FOLFOX is allowed. Dose modifications are allowed, but all 3 cycles must have been completed.
3. Must have undergone a surgical resection with definitive intent, either by open or laparoscopic resection of the primary gastric or GE junction cancer. Patients must have undergone a total gastrectomy, subtotal gastrectomy, or distal gastrectomy (depending on the location of primary gastric lesion) with at least a modified D2 lymphadenectomy.
4. Must be deemed as a good candidate for adjuvant chemotherapy or chemoradiation (to start within 3 months of surgery), in the opinion of the treating investigator. Plan must be to start adjuvant therapy within 90 days of surgery; adjuvant treatment cannot begin more than 90 days after surgery.
5. Must have diagnostic biopsy tissue (pre-neoadjuvant chemo) available for genetic testing.
6. Must have surgical tissue (post-neoadjuvant chemo) available for genetic testing.
7. Must be > 18 years of age.
8. Must be able to provide informed consent.
9. Must have adequate kidney, liver, and bone marrow function, within 28 days prior to registration, as follows:

   i. Hemoglobin ≥ 8.0 gm/dL

   ii. Absolute neutrophil count (ANC) ≥ 1500 cells/mm3

   iii. Platelet count ≥ 75,000 /mm3

   iv. Calculated creatinine clearance of > 60 mL/min/m2, calculated as follows:

   For males = ((140 - age [years]) x (body weight [kg])) / ((72) x (serum creatinine [mg/dL])

   For females = 0.85 x male value

   v.Total bilirubin ≤ 1.5 times upper limit of normal (ULN)

   vi.AST (aspartate aminotransferase) (SGOT) and ALT (alanine transaminase) (SGPT) ≤ 3.0 times the ULN
10. Must have life expectancy of greater than 3 months.
11. Must have an ECOG (Eastern Cooperative Oncology Group) performance status 0-2.
12. Male or female patients of childbearing potential must be willing to use contraceptive precautions throughout the trial and 3 months following discontinuation of study treatment. Post-menopausal women must be amenorrheic for at least 12 months to be considered of non-childbearing potential.

Exclusion Criteria:

1. Other than the 3 cycles of neoadjuvant chemotherapy and surgery (mentioned above), must not have received other treatment for their gastric cancer.
2. Female patients who are pregnant, breast feeding, or of childbearing potential without a negative pregnancy test prior to baseline. Women of childbearing potential must have a negative serum pregnancy test as a part of eligibility, within 28 days of registration.
3. Patients unwilling or unable to comply with the protocol, or provide informed consent.
4. Patients with clinical evidence of metastatic disease.
5. Any medical condition that, in the opinion of the investigator, would exclude the patient from participating in this study and treatment plan.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2018-06-22 (Actual); Primary Completion 2020-03-17 (Actual); Study Completion 2020-06-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tannaz Armaghany, MD, Principal Investigator — Baylor College of Medicine
Locations (4):
- United States (4):
  - Baylor College of Medicine Medical Center - McNair Campus, Houston, Texas
  - Baylor College of Medicine, Houston, Texas
  - Baylor St. Lukes Medical Center, Houston, Texas
  - Harris Health System- Smith Clinic, Houston, Texas

REFERENCES:
- [Background] Cunningham D, Allum WH, Stenning SP, Thompson JN, Van de Velde CJ, Nicolson M, Scarffe JH, Lofts FJ, Falk SJ, Iveson TJ, Smith DB, Langley RE, Verma M, Weeden S, Chua YJ, MAGIC Trial Participants. Perioperative chemotherapy versus surgery alone for resectable gastroesophageal cancer. N Engl J Med. 2006 Jul 6;355(1):11-20. doi: 10.1056/NEJMoa055531. PMID 16822992
- [Background] Macdonald JS, Smalley SR, Benedetti J, Hundahl SA, Estes NC, Stemmermann GN, Haller DG, Ajani JA, Gunderson LL, Jessup JM, Martenson JA. Chemoradiotherapy after surgery compared with surgery alone for adenocarcinoma of the stomach or gastroesophageal junction. N Engl J Med. 2001 Sep 6;345(10):725-30. doi: 10.1056/NEJMoa010187. PMID 11547741
- [Background] Cunningham D, Starling N, Rao S, Iveson T, Nicolson M, Coxon F, Middleton G, Daniel F, Oates J, Norman AR; Upper Gastrointestinal Clinical Studies Group of the National Cancer Research Institute of the United Kingdom. Capecitabine and oxaliplatin for advanced esophagogastric cancer. N Engl J Med. 2008 Jan 3;358(1):36-46. doi: 10.1056/NEJMoa073149. PMID 18172173
- [Background] Ychou M, Boige V, Pignon JP, Conroy T, Bouche O, Lebreton G, Ducourtieux M, Bedenne L, Fabre JM, Saint-Aubert B, Geneve J, Lasser P, Rougier P. Perioperative chemotherapy compared with surgery alone for resectable gastroesophageal adenocarcinoma: an FNCLCC and FFCD multicenter phase III trial. J Clin Oncol. 2011 May 1;29(13):1715-21. doi: 10.1200/JCO.2010.33.0597. Epub 2011 Mar 28. PMID 21444866
- [Background] Enzinger PC, Burtness BA, Niedzwiecki D, Ye X, Douglas K, Ilson DH, Villaflor VM, Cohen SJ, Mayer RJ, Venook A, Benson AB 3rd, Goldberg RM. CALGB 80403 (Alliance)/E1206: A Randomized Phase II Study of Three Chemotherapy Regimens Plus Cetuximab in Metastatic Esophageal and Gastroesophageal Junction Cancers. J Clin Oncol. 2016 Aug 10;34(23):2736-42. doi: 10.1200/JCO.2015.65.5092. Epub 2016 Jul 5. PMID 27382098
- [Background] Dikken JL, van Sandick JW, Maurits Swellengrebel HA, Lind PA, Putter H, Jansen EP, Boot H, van Grieken NC, van de Velde CJ, Verheij M, Cats A. Neo-adjuvant chemotherapy followed by surgery and chemotherapy or by surgery and chemoradiotherapy for patients with resectable gastric cancer (CRITICS). BMC Cancer. 2011 Aug 2;11:329. doi: 10.1186/1471-2407-11-329. PMID 21810227
- [Background] Smyth EC, Fassan M, Cunningham D, Allum WH, Okines AF, Lampis A, Hahne JC, Rugge M, Peckitt C, Nankivell M, Langley R, Ghidini M, Braconi C, Wotherspoon A, Grabsch HI, Valeri N. Effect of Pathologic Tumor Response and Nodal Status on Survival in the Medical Research Council Adjuvant Gastric Infusional Chemotherapy Trial. J Clin Oncol. 2016 Aug 10;34(23):2721-7. doi: 10.1200/JCO.2015.65.7692. Epub 2016 Jun 13. PMID 27298411
- [Background] Lee J, Lim DH, Kim S, Park SH, Park JO, Park YS, Lim HY, Choi MG, Sohn TS, Noh JH, Bae JM, Ahn YC, Sohn I, Jung SH, Park CK, Kim KM, Kang WK. Phase III trial comparing capecitabine plus cisplatin versus capecitabine plus cisplatin with concurrent capecitabine radiotherapy in completely resected gastric cancer with D2 lymph node dissection: the ARTIST trial. J Clin Oncol. 2012 Jan 20;30(3):268-73. doi: 10.1200/JCO.2011.39.1953. Epub 2011 Dec 19. PMID 22184384
- [Background] Park SH, Sohn TS, Lee J, Lim DH, Hong ME, Kim KM, Sohn I, Jung SH, Choi MG, Lee JH, Bae JM, Kim S, Kim ST, Park JO, Park YS, Lim HY, Kang WK. Phase III Trial to Compare Adjuvant Chemotherapy With Capecitabine and Cisplatin Versus Concurrent Chemoradiotherapy in Gastric Cancer: Final Report of the Adjuvant Chemoradiotherapy in Stomach Tumors Trial, Including Survival and Subset Analyses. J Clin Oncol. 2015 Oct 1;33(28):3130-6. doi: 10.1200/JCO.2014.58.3930. Epub 2015 Jan 5. PMID 25559811

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm 1: Adjuvant Chemotherapy | Arm 2: Adjuvant Chemoradiation
Started | 4 | 2
Completed | 3 | 2
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1: Adjuvant Chemotherapy | Arm 2: Adjuvant Chemoradiation | Total
Number analyzed (Participants) | 4 | 2 | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.9 (12.6) | 38.5 (6.2) | 51.4 (14.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 2 | 0 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 2 | 5
  Not Hispanic or Latino | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 3 | 2 | 5
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
ECOG performance status [Count of Participants; unit: Participants] — The Eastern Cooperative Oncology Group (ECOG) performance score is a scale to assess how the disease affects the daily living abilities of the patient. ECOG score ranges from 0 to 5, with 0 denoting perfect health and 5 death. Less ECOG score is considered better living ability.
  ECOG 0:Fully active, able to carry on all pre-disease performance without restriction ECOG 1:Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work
  Participants
    ECOG score 0 | 3 | 2 | 5
    ECOG score 1 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Complete the Recommended Therapy From Each Arm
Description: The number of patients who complete the recommended therapy will be counted for each arm.
Time Frame: From date of assigned therapy up to 17 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: Adjuvant Chemotherapy | Arm 2: Adjuvant Chemoradiation
Number analyzed (Participants) | 4 | 2
Participants | 3 | 2

2. Secondary Outcome: Median Time to Recurrence
Description: Disease recurrence will be defined as radiographic tumor evidence detected by surveillance imaging. Confirmation of recurrence by biopsy will be at the discretion of the treating physician. This study closed early on June 18, 2020. It was earlier than one planned because of the lack of accrual.
Time Frame: From the end of completion of assigned therapy, subjects undergo follow-up every 3 months for a total of 36 months(planned) after the date of surgery or until the study closure
Population: All patients who are enrolled on the study and begin any of their intended post-operative adjuvant therapy will be counted as evaluable for the study. This inclusion will be regardless of how much of the postoperative treatment they ultimately receive.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm 1: Adjuvant Chemotherapy | Arm 2: Adjuvant Chemoradiation
Number analyzed (Participants) | 4 | 2
months | NA [5.96 to NA] — The median recurrence time was NA therefore the upper 95% confidence interval is NA. | NA [NA to NA] — There was no recurrence occurred during the time period we observed. Therefore, the recurrence has not been reached to the median.

ADVERSE EVENTS:
Time Frame: From the end of completion of assigned therapy, subjects undergo follow-up every 3 months for a total of 36 months(planned) after the date of surgery or until the study closure
Arm/Group | Arm 1: Adjuvant Chemotherapy | Arm 2: Adjuvant Chemoradiation
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/4 | 1/2
Other Adverse Events (participants affected / at risk) | 3/4 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1: Adjuvant Chemotherapy (N=4) | Arm 2: Adjuvant Chemoradiation (N=2)
Gastrointestinal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1: Adjuvant Chemotherapy (N=4) | Arm 2: Adjuvant Chemoradiation (N=2)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (2)
Vomiting (Gastrointestinal disorders) | 2 (2) | 2 (2)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 2 (2) | 2 (2)
General disorders and administration site conditions - Other, specify (General disorders) | 0 (0) | 1 (1) — This adverse event was monitored/assessed without regard to the specific Adverse Event Term.
Pain (General disorders) | 0 (0) | 2 (2)
Upper respiratory infection (Infections and infestations) | 0 (0) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Alkaline phosphatase increased (Investigations) | 1 (1) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 1 (1)
Lymphocyte count decreased (Investigations) | 1 (1) | 2 (2)
Neutrophil count decreased (Investigations) | 1 (1) | 1 (1)
Platelet count decreased (Investigations) | 1 (1) | 1 (1)
Weight loss (Investigations) | 1 (1) | 0 (0)
White blood cell decreased (Investigations) | 0 (0) | 2 (2)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-01-29): https://cdn.clinicaltrials.gov/large-docs/41/NCT03515941/Prot_SAP_000.pdf